CLINICAL TRIAL: NCT03426423
Title: Assessing the Efficacy and Impact of a Personalized Smoking Cessation Intervention Among Type 2 Diabetic Smokers in a Randomized Controlled Trial
Brief Title: Diabetes and Smoking Cessation: a Gender-Oriented Study
Acronym: DiSCGO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment rate too low (COVID-19 pandemic), end of funding
Sponsor: Carole Clair (Other)
Responsible Party: Sponsor-Investigator, Carole Clair, Principal Investigator, Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland
Organization: Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2017-00812
Record Dates: First submitted 2018-01-18; First posted 2018-02-08 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Smoking Cessation; Diabetes Type 2
Keywords: Gender; Metabolism; Microbiota
MeSH Terms: conditions — Smoking Cessation; Diabetes Mellitus, Type 2; Coitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: According to the article 18 of the LRH, participants will not be given the full information regarding the main purpose of the study (assess the efficacy of a smoking cessation trial) in order not to influence participants regarding the intervention and also to decrease selection bias (only smokers motivated to quit would take part and thus induce a selection bias). Methodologically, such a blinding to procedure would allow a better assessment of its efficacy. Furthermore, risks associated to the intervention are considered as very low. Participants will be informed a posteriori once they have completed the study or before in case they remove their consent or quit the study.
  The outcome assessor will be a research collaborator independent of the study nurse who performed the intervention and blinded to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 12 weeks smoking cessation intervention tailored to diabetic and gender specificities, delivered by a study nurse.
  Interventions: Other: Behavioral smoking cessation intervention
- Control (Active Comparator): Usual care comprising a unique intervention of 5-10 minutes, non tailored smoking cessation intervention, delivered by a study nurse.
  Interventions: Other: Control

INTERVENTIONS:
Other: Behavioral smoking cessation intervention — The intervention consists in a behavioral smoking cessation intervention combined with pharmacotherapy. The intervention is tailored it to specificities of participants based on findings from the previous phase of our study (DISCGO-MIX, Swissethics ID PB_2016-01459).
  Counseling will cover topics such as assessing ambivalence and enhancing motivation with motivational interviewing methods, identifying barriers to quit, coping with cravings and intensive relapse prevention strategies. Participants will be advised to use over the counter nicotine replacement bi-therapy (NTR). A 2-week starting kit, consisting of nicotine transdermal patch and a short acting NRT (lozenge, gums, inhaler or mouth spray) will be provided to participants for free, if they wish to take NRT.
  The behavioral intervention will last 30-45 minutes, and will be conducted by a research nurse using an interview guide.
  Arms: Intervention
Other: Control — Participants assigned to the control group will receive a less intensive and non-tailored intervention for smoking cessation.
  For this arm the structured 3 steps AAR approach will be used:
  Ask for smoking status. Advise to quit in a clear manner. Refer to external help: participants will receive a booklet with information on smoking cessation (non specific to diabetes and gender) and links to support facilities (national quitline, smoking cessation clinic, websites, self-help).
  This unique intervention of 5-10 minutes will be performed by the research nurse.
  Arms: Control

SUMMARY:
People with diabetes still smoke at equivalent rates as non-diabetics. There is lack of evidence regarding interventions for smoking cessation among individuals with diabetes. The aim of this project is to assess the 12 months efficacy of a smoking cessation intervention tailored to diabetes and gender specificities, in a population of 500 smokers with type 2 diabetes. The secondary objectives are to assess the impact of smoking cessation on anthropometric outcomes, diabetes control and renal function and fecal microbiota.

DETAILED DESCRIPTION:
Smoking and diabetes are both major public health burden. They act synergistically on morbidity and mortality. Micro and macro-vascular complications are dramatically increased among diabetic smokers; however people with diabetes still smoke at equivalent rates as non-diabetics. There is lack of evidence regarding interventions for smoking cessation among individuals with diabetes and the small number of existent studies has yielded mixed results.

The aim of this project is to assess the 52 weeks (12 months) efficacy of a smoking cessation intervention tailored to diabetes and gender specificities, in a population of smokers with type 2 diabetes.

The secondary objectives are to assess the impact of smoking cessation on anthropometric outcomes, diabetes control and renal function.

The exploratory objectives are to assess the impact of smoking cessation on fecal microbiota The nested sub-study's exploratory objectives are to explore the associations between social stigma and diabetes, and mental health and diabetes.

The study design is an open label, randomized controlled trial with a nested cross-sectional study.

Participants will be recruited from the Policlinique Médicale Universitaire (PMU) of Lausanne, the university hospital in Lausanne (CHUV) and peripheral hospitals, private practices of general internists and specialists of diabetology and the community.

All screening procedures will be performed by a study nurse delegated by the PI based at the PMU. Eligible participants will be randomly allocated to either the intervention or control arm. Stratified randomization by sex will be done to ensure that the proportion of men and women is the same in both arms. Demographic data, medical data and specific questionnaires related to diabetes, smoking, gender and mental health /social stigma will be administered at baseline and a blood sample will be taken. In a subsample of 80 selected participants change in microbiota in stool will be measured at baseline, 3, 8 and 26 weeks after smoking cessation (or after baseline for continuing smokers).The intervention group will have 4 individual counseling sessions over 12 weeks. The control group will have 1 counseling session and will be given written information on smoking cessation. The control group will receive 2 telephone calls at 3 weeks and 8 weeks and a control visit at 12 weeks to assess smoking cessation (without counseling). Both groups will have a follow-up visit at 26 weeks and at 52 weeks.

500 participants in total will be included, 250 in each intervention arm. The duration of the study is planned for 3 years ( 4-5 participants/week during 2 years and follow-up of 52 weeks).

For the main outcome the analyses will be performed intention to treat. Participants lost to follow-up will be considered as smokers. The primary outcome (52 weeks smoking abstinence) will be compared using Pearson's chi-squared tests.

Power calculations indicate that a sample size of approximately 400 people is needed to detect a 10% difference in smoking abstinence between intervention and control groups (52 weeks continuous smoking abstinence equal to 0.2 in the intervention group and 0.1 in the control group) with a two-sample proportions test using Pearson's chi-squared test, power 80%, significance level 0.05. With an expected 20% attrition rate, the sample will be increased to 500 participants.

This study will be conducted in compliance with the protocol, the current version of the Declaration of Helsinki, the ICH-GCP as well as all national legal and regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature;
* Having smoked > 100 cigarettes during his/her entire life and currently smoking cigarettes (no minimal threshold);
* Having been diagnosed with a type 2 diabetes;
* Being ≥ 18 years old;
* Speaking and understanding French

Exclusion Criteria:

* Not being able to give an informed consent and follow the procedure of the study (due to dementia, psychological disorder, language problem);
* Being pregnant or breastfeeding;
* Being enrolled in another smoking cessation study or program or in a multi-behavioral program including smoking cessation;
* Enrolment of the investigator or other research collaborators, their family members, employees and other dependent persons;
* Planning to move out of Switzerland within the next year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Identification is based on self-representation of gender eligibility with the possibility to self identify as transgender.
Enrollment: 48 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Continuous smoking abstinence | Measured at 52 weeks
  continuous abstinence rate from week 12 (end of intervention) to week 52 (end of follow-up), defined as self-report of no smoking or use of other nicotine containing products (ENDS, smokeless tobacco) since the previous visit or contact, confirmed by expired monoxide level < 10 ppm.

SECONDARY OUTCOMES:
Point prevalence smoking abstinence | Change is measured at 12 week
  7-day point-prevalence abstinence validated by CO
Point prevalence smoking abstinence | Change is measured at 26 weeks
  7-day point-prevalence abstinence validated by CO
Point prevalence smoking abstinence | Change is measured at 52 weeks
  7-day point-prevalence abstinence validated by CO
Motivation to quit smoking | Change is measured from baseline to 12 week
  Change in motivation to quit (according to Prochaska and Di Clemente)
Motivation to quit smoking | Change is measured from baseline to 26 week
  Change in motivation to quit (according to Prochaska and Di Clemente)
Motivation to quit smoking | Change is measured from baseline to 52 week
  Change in motivation to quit (according to Prochaska and Di Clemente)
Harm reduction | Change is measured at 26 week
  Decrease in ≥ 50% of cigarette consumption
Harm reduction | Change is measured at 52 week
  Decrease in ≥ 50% of cigarette consumption
Weight change | Change from baseline to 26 week
  Change in body weight measured in kg
Weight change | Change from baseline to 52 week
  Change in body weight measured in kg
Metabolic control | Change is measured from baseline to 12 week
  Change in HbA1c
Metabolic control | Change is measured from baseline to 26 week
  Change in HbA1c
Metabolic control | Change is measured from baseline to 52 week
  Change in HbA1c
Renal function | Change is measured from baseline to 3 weeks.
  Change in renal function represented by eGFR and albumin/creatinine ratio
Renal function | Change is measured from baseline to 8 weeks.
  Change in renal function represented by eGFR and albumin/creatinine ratio
Renal function | Change is measured from baseline to 26 weeks.
  Change in renal function represented by eGFR and albumin/creatinine ratio
Number of smoking quit attemps | Change is measured from baseline to 12 week
  Number of quit attemps defined as smoking abstinence > 24h
Number of smoking quit attempts | Change is measured from baseline to 26 week
  Number of quit attempts defined as smoking abstinence > 24h
Number of smoking quit attempts | Change is measured from baseline to 52 week.
  Number of quit attempts defined as smoking abstinence > 24h
Change in waist circumference | Change from baseline to 26 week
  Change in waist circumference in cm
Change in waist circumference | Change from baseline to 52 week.
  Change in waist circumference in cm
Continuous smoking abstinence | At week 12
  continuous abstinence rate from baseline to week 12, defined as self-report of no smoking or use of other nicotine containing products (ENDS, smokeless tobacco) since the previous visit or contact, confirmed by expired monoxide level < 10 ppm.
Continuous smoking abstinence | At week 26
  continuous abstinence rate from week 12 to week 26, defined as self-report of no smoking or use of other nicotine containing products (ENDS, smokeless tobacco) since the previous visit or contact, confirmed by expired monoxide level < 10 ppm.

OTHER OUTCOMES:
Exploratory microbiota outcome | Change is measured from baseline to 4 weeks.
  Change in fecal microbiota
Exploratory microbiota outcome | Change is measured from baseline to 8 weeks.
  Change in fecal microbiota
Exploratory microbiota outcome | Change is measured from baseline to 26 weeks.
  Change in fecal microbiota

CONTACTS AND LOCATIONS:
Overall Officials: Carole Clair, MD, MSc, Principal Investigator — Center for Primary Care and Public Health, Lausanne University
Locations (1):
- Center for Primary Care and Public Health, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clair C, Augsburger A, Birrer P, Locatelli I, Schwarz J, Greub G, Zanchi A, Jacot-Sadowski I, Puder JJ. Assessing the efficacy and impact of a personalised smoking cessation intervention among type 2 diabetic smokers: study protocol for an open-label randomised controlled trial (DISCGO-RCT). BMJ Open. 2020 Nov 19;10(11):e040117. doi: 10.1136/bmjopen-2020-040117. PMID 33444198